CLINICAL TRIAL: NCT03250364
Title: Compression Bandages in Upper Limb Lymphedema After Breast Cancer
Brief Title: Compression Bandages in Upper Limb Lymphedema
Acronym: CB-ULL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18/2010
Record Dates: First submitted 2017-08-04; First posted 2017-08-15 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: 5 goups: Multilayer bandage group; Double compression bandage group; Cohesive bandage group; Adhesive compression bandage group; Kinesiotaping bandage group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Multilayer bandage group (Experimental): Manual lymphatic drainage (MLD) + upper limb (UL) exercises + educational strategy + multilayer bandage consisting of three layers. The first was a 100% cotton tubular bandage which will be directly placed on the skin to prevent any injury ("Tubinylex TM"). The second layer is a paddle with the purpose of unify and increase pressure (Emulsified Latex FoamTM 8mm, Thuasne, France); and the third layer of inelastic bandages (6, 8 and/or 10 cm Rosidal K Short Stretch Bandage, Germany). All the bandage layers will be placed from caudal to cranial in a circular disposition, overlapping in one third the previous layer for a correctly cover of the limb and not to leave open spaces. The cotton tubular bandage and the short-stretch bandage could be cleaned without losing their material properties.
  Interventions: Device: Multilayer bandage; Other: Manual lymphatic drainage (MLD) + Intermittent Pneumatic Compression; Other: Upper limb exercises; Behavioral: Educational strategy
- Simplified multilayer bandage group (Experimental): Manual lymphatic drainage (MLD) + upper limb (UL) exercises + educational strategy + double compression bandage consisting of two layers, made up of a first rigid cotton bandage (11 cm Bande coton Short Stretch; Thuasne, France) and a second elastic bandage ("BiflexTM" 16 light; Thuasne, France). The two layers will be placed caudal to cranial in a circular manner, overlapping in one third the previous layer. The elastic bandage have squares drawn to help to the physiotherapist to control the stretch they given to the bandage. The two bandages could be cleaning without losing their properties. If there was any oedema concentration or a fibrous place, a paddle pad will be put in these places ("Mobiderm TM", Thuasne, France).
  Interventions: Device: Double compression bandage; Other: Manual lymphatic drainage (MLD) + Intermittent Pneumatic Compression; Other: Upper limb exercises; Behavioral: Educational strategy
- Cohesive bandage group (Experimental): Manual lymphatic drainage (MLD) + upper limb (UL) exercises + educational strategy + cohesive bandage consisting of a single short-stretched layer that will be put directly on the subject skin and stick on itself (10cm 3M CobanTM Minnesota Mining and Manufacturing Co, United States). It will be placed in a circular manner distal to cranial with a paddle pad in the elbow fold not to damage this moving part. This bandage will be reused twice in the same subject.
  Interventions: Device: Cohesive bandage; Other: Manual lymphatic drainage (MLD) + Intermittent Pneumatic Compression; Other: Upper limb exercises; Behavioral: Educational strategy
- Adhesive compression bandage group (Experimental): Manual lymphatic drainage (MLD) + upper limb (UL) exercises + educational strategy + adhesive compression bandage consisting of an elastic bandage ("BiplastTM" Thuasne, France. Measures: 10cm x 2,5 m) which will put over a pre-tape bandage not to damage the skin. It will be placed in a circular disposition from distal to cranial. In each physiotherapy session, the bandage has to be replaced with a new one.
  Interventions: Device: Adhesive compression bandage; Other: Manual lymphatic drainage (MLD) + Intermittent Pneumatic Compression; Other: Upper limb exercises; Behavioral: Educational strategy
- Kinesiotaping bandage group (Experimental): Manual lymphatic drainage (MLD) + upper limb (UL) exercises + educational strategy + kinesiotaping bandage consisting of K-Active" Tape. The k-tape will be pasted directly on the skin and put longitudinally in thin bands in a cranio-caudal disposition. The width of the bandage will be of 5cm, and will be cut in four bands that will cover all the upper limb cranial to caudal in a spiral way surrounded it. The bandage will be placed moving the limb into internal and external rotation for putting the skin in a little stretch without lengthen the tape.
  Interventions: Device: Kinesiotaping bandage; Other: Manual lymphatic drainage (MLD) + Intermittent Pneumatic Compression; Other: Upper limb exercises; Behavioral: Educational strategy

INTERVENTIONS:
Device: Multilayer bandage — See arm/group descriptions
  Arms: Multilayer bandage group
Device: Double compression bandage — See arm/group descriptions
  Arms: Simplified multilayer bandage group
Device: Cohesive bandage — See arm/group descriptions
  Arms: Cohesive bandage group
Device: Adhesive compression bandage — See arm/group descriptions
  Arms: Adhesive compression bandage group
Device: Kinesiotaping bandage — See arm/group descriptions
  Arms: Kinesiotaping bandage group
Other: Manual lymphatic drainage (MLD) + Intermittent Pneumatic Compression — MLD using a modification of the strokes described by Leduc will be applied to lymphedema "resorption". It will be included resorption maneuver in the oedematous areas of the affected limb, in cranial to caudal direction, since the physiotherapist seeing a change in the tissue qualities of the oedema. Then, the subjects will be received thirty minutes of Intermittent Pneumatic Compression ("EureducTM") with a pression of 40 mmHg.
Other: Upper limb exercises — After the bandage will be put, proprioceptive neuromuscular facilitation exercises without resistance in two diagonal in asymmetrical reciprocal patterns with the affected limb will be taught. The first diagonal into flexion from hitch hike to swat fly, and into extension from swat fly to hitch hike, and the second diagonal from hand in opposite pocket to carry tray, and into extension from carry tray to hand in opposite pocket. These exercises must be done at home two times per day, ten repetitions each exercise.
Behavioral: Educational strategy — Instructions about lymphatic system anatomy and pato-physiology, the prevention and identification of possible lymphedema complication or infection, how to use and exercise this arm, avoidance of trauma, injury, an excess of heat and arm constriction.

SUMMARY:
Despite different types of bandages are using in the lymphedema treatment, numerous of them have not been directly compared. The aim of this study is to compare the efficacy of five different kinds of bandages on limb volume and lymphedema-related symptoms. It was also measured as secondary variables the comfort of the bandage related by the participants and the directly cost of each kind of bandage during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women after breast cancer surgery undergoing upper limb lymphedema not previously treated
* Having more than two centimeters between two adjacent measurements between the lymphedematous and the contralateral upper limb
* The presence of heaviness, tension or fovea in the affected limb
* More than six months post-surgery or radiation to eliminate the possibility of being a post-chirurgical oedema

Exclusion criteria will be:

* Bilateral breast cancer surgery
* Only hand lymphedema
* Active cutaneous infection
* A loco-regional cancer recurrence
* The impossibility of complete all the physical therapy sessions
* A primary lymphedema
* Women with lymphedema symptoms like thickness and heaviness in the upper limb but without a difference of two centimeters in two adjacent points
* Any contraindication to physiotherapy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Change in arm volume | 3 assessments to evaluate changes: at baseline (before intervention), after intervention (1 month from baseline) and 6 months after intervention
  To assess the volume of the limb it will be used the circumference measurement. The assessment will be with the subject in upright position with the arm placed on a table, the forearm relaxed on the table, the shoulder in a neutral rotation, a flexion of 45º of the elbow, and forearms in supine position. The reference will be the elbow fold where was measure the circumference of the limb in 5cm intervals. The circumference measurements will be converted into volume values with the truncated cone formula in each 5 centimeters long.
Change in heath related quality of life lymphedema | 3 assessments to evaluate changes: at baseline (before intervention), after intervention (1 month from baseline) and 6 months after intervention
  It will be assessed by Lymphedema specific PRO instrument: Upper Limb Lymphedema (ULL)27 spanish validated version

SECONDARY OUTCOMES:
Change in comfort of the bandage | 3 assessments to evaluate changes: at baseline (before intervention), after intervention (1 month from baseline) and 6 months after intervention
  Numeric scale ranging from 0-10: 0 comfortable - 10: very uncomfortable

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Physiotherapy in women´s health research group. University of Alcalà, Alcalà de Henares, Madrid
  - University of Alcalá. FPSM research group. HUPA, Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: No